CLINICAL TRIAL: NCT03451422
Title: A Randomized, Double-blind, Placebo-controlled Phase 1b Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Multiple Ascending Subcutaneous Doses of Efavaleukin Alfa in Subjects With Systemic Lupus Erythematosus
Brief Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of Efavaleukin Alfa in Participants With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 20170103; 2017-002564-40 (EudraCT Number)
Record Dates: First submitted 2018-02-01; First posted 2018-03-01 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Efavaleukin Alfa; Systemic lupus erythematosus; Phase 1b
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Intervention Model Description: This phase 1b study is a double-blind, placebo controlled multiple ascending dose (MAD) study to evaluate the safety and tolerability of Efavaleukin Alfa in participants with systemic lupus erythematosus (SLE) and to determine the recommended phase 2 dose(s). Participants will be treated for a total of 12 weeks followed by a 6 week follow-up period. Five dosing cohorts are planned for the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Efavaleukin Alfa (Experimental): Approximately 29 participants will be randomized in a 5:2 ratio (cohorts 1, 2, and 3) or in a 3:1 ratio (cohorts 4 and 5) to Efavaleukin Alfa or placebo in addition to standard of care therapy. Efavaleukin Alfa or placebo will be administered either weekly (QW) or biweekly (Q2W).
  Interventions: Drug: Efavaleukin Alfa
- Placebo (Placebo Comparator): Approximately 29 participants will be randomized in a 5:2 ratio (cohorts 1, 2, and 3) or in a 3:1 ratio (cohorts 4 and 5) to Efavaleukin Alfa or placebo in addition to standard of care therapy. Efavaleukin Alfa or placebo will be administered either weekly (QW) or biweekly (Q2W).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efavaleukin Alfa — Efavaleukin Alfa will be administered by subcutaneous (SC) injection in the abdomen, thigh or upper arm.
  Arms: Efavaleukin Alfa
Drug: Placebo — The placebo will be administered by subcutaneous (SC) injection in the abdomen, thigh or upper arm.
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of subcutaneous (SC) dose administrations of Efavaleukin Alfa in participants with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Age ≥ 18 years to ≤ 70 years at screening.
* Fulfills diagnostic criteria for SLE according to the Systemic Lupus International Collaborating Clinics (SLICC) criteria or by at least 4 of the 11 criteria of the 1997 American College of Rheumatology (ACR) classification criteria for SLE, with a history of at least one of the following:

  * Antinuclear antibody ≥ 1:80; or
  * Elevated anti-dsDNA antibodies
* May be taking ≤ 3 systemic SLE treatments and the dose must be stable for ≥ 4 weeks prior to day 1.
* Prednisone dose ≤ 20 mg daily (or other equivalent oral corticosteroid) with stable dose ≥ 2 weeks prior to day 1.
* Normal or clinically acceptable ECG values (12-lead reporting ventricular rate and PR, QRS, QT and QTc interval) at screening and baseline based on opinion of the investigator.
* Immunizations (tetanus, diphtheria, pertussis [Td/Tdap]), seasonal influenza (during flu season), and pneumococcal (polysaccharide) vaccinations] up to date per local standards as determined by the investigator.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply.

Disease Related

- History of lupus nephritis requiring induction therapy and/or lupus cerebritis ≤ 1 year prior to screening.

Other Medical Conditions

* Diagnosis of inflammatory joint or skin disease other than SLE which would interfere with SLE disease assessment based on investigator judgement.
* Diagnosis of fibromyalgia which would interfere with SLE assessment according to the investigator.
* Prosthetic joint infection within 3 years of screening or native joint infection within 1 year prior to screening.
* Active infection (including chronic or localized infections) for which anti-infectives were indicated within 4 weeks prior to day 1 OR presence of serious infection, defined as requiring hospitalization or intravenous anti-infectives within 8 weeks prior to day 1.
* Known history of active tuberculosis.
* Positive test for tuberculosis during screening defined as either:

  * positive purified protein derivative (PPD) (≥ 5 mm of induration at 48 to 72 hours after test is placed) OR positive Quantiferon test
* a positive PPD and a history of Bacillus Calmette-Guérin vaccination are allowed with a negative Quantiferon test and negative chest X-ray.

  * a positive PPD test (without a history of Bacillus Calmette-Guérin vaccination) or a positive or indeterminate Quantiferon test are allowed if they have ALL of the following at screening:
* no symptoms per tuberculosis worksheet provided by Amgen
* documented history of a completed course of adequate prophylaxis (completed treatment for latent tuberculosis per local standard of care prior to the start of investigational product)
* no known exposure to a case of active tuberculosis after most recent prophylaxis
* negative chest X-ray.
* Positive for hepatitis B surface antigen, hepatitis B core antibody (confirmed by hepatitis B DNA polymerase chain reaction [PCR] test) or detectable hepatitis C virus RNA by PCR (screening is generally done by hepatitis C antibody [HepCAb], followed by hepatitis C virus RNA by PCR if HepCAb is positive). A history of hepatitis B vaccination without history of hepatitis B is allowed.
* Positive for Human Immunodeficiency Virus (HIV) at screening, or known to be HIV positive.
* Presence of one or more significant concurrent medical conditions per investigator judgment, including but not limited to the following:

  * poorly controlled diabetes or hypertension
  * chronic kidney disease stage IIIb, IV, or V
  * symptomatic heart failure (New York Heart Association class II, III, or IV)
  * myocardial infarction or unstable angina pectoris within the past 12 months prior to randomization
  * severe chronic pulmonary disease (eg, requiring oxygen therapy)
  * multiple sclerosis or any other demyelinating disease
  * major chronic inflammatory disease or connective tissue disease other than SLE (eg, RA).
* Malignancy except non-melanoma skin cancers, cervical or breast ductal carcinoma in situ within 5 years of screening.
* Participants with a urine test positive for illicit drugs or alcohol at the screening visit. Prescription medications detected by the drug test are allowed if they are being taken under the direction of a physician.
* History of alcohol or substance abuse within 6 months of screening.
* Current smoker, and/or use of any nicotine or tobacco containing products within the last 6 months prior to day 1. These types of products include but are not limited to: snuff, chewing tobacco, cigars, cigarettes, electronic cigarettes, pipes, or nicotine patches.
* Participant unwilling to limit alcohol consumption to ≤ 1 drink of alcohol per day and ≤3 drinks per week for the duration of the study, where a drink is equivalent to 12 ounces of regular beer, 8 to 9 ounces of malt liquor, 5 ounces of wine, or 1.5 ounces of 80 proof distilled spirits.

Prior/Concomitant Therapy

* Currently receiving or had treatment with: cyclophosphamide, chlorambucil, nitrogen mustard, or any other alkylating agent ≤ 6 months prior to day 1 OR oral calcineurin inhibitors (eg, cyclosporine, tacrolimus, sirolimus) ≤ 4 weeks prior to day 1.
* Current or previous treatment for SLE with a biologic agent as follows: rituximab < 6 months prior to day 1, belimumab < 3 months prior to day 1, abatacept < 8 weeks prior to day 1.
* Currently receiving or had treatment with T cell depleting agents (eg, antithymocyte globulin, Campath) or recombinant IL-2 (eg, Proleukin).
* Participants who have received intra-articular or systemic corticosteroid injections within 4 weeks prior to day 1 or topical steroids within 2 weeks prior to day 1.
* Administration of herbal supplements, vitamins, or nutritional supplements within 30 days prior to the first dose of investigational product, and continuing use, if applicable, will be reviewed by the Investigator and the Amgen Medical Monitor to determine acceptability. Written documentation of this review and Amgen acknowledgment is required for participant participation.

Prior/Concurrent Clinical Study Experience

* Currently receiving treatment in another investigational device or drug study, or less than 30 days at day 1 since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Participant previously enrolled in this study may not be re-enrolled unless they fulfill the following criteria:

  * Have completed the study previously without any adverse events deemed related to study drug.
  * Have received the last dose of Efavaleukin Alfa/placebo > 6 months prior to the screening visit.
  * Must not have tested positive for neutralizing antibodies against Efavaleukin Alfa at any time.

Diagnostic Assessments

* Presence of laboratory abnormalities at screening including the following:

  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 1.5x upper limit of normal (ULN)
  * Serum total bilirubin (TBL) ≥ 1.5 mg/dL (≥ 26 μmol/L)
  * Hemoglobin < 9.0 g/dL(< 90 g/L)
  * Platelet count < 100,000/mm^3 (100 x 10^9/L)
  * White blood cell count < 2,000 cells/mm^3 (2.0 x 10^9/L)
  * Absolute neutrophil count (ANC) < 1,000/mm^3 (1.0 x 10^9/L)
  * Calculated glomerular filtration rate of ≤ 50 mL/min/1.73 m^2 using the Modification of Diet in Renal Disease (MDRD) formula.
* Any other laboratory abnormality, which, in the opinion of the investigator, poses a safety risk, will prevent the participant from completing the study, will interfere with the interpretation of the study results, or might cause the study to be detrimental to the participant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (15):
- United States (6):
  - Pinnacle Research Group LLC, Anniston, Alabama
  - Wallace Rheumatic Studies Center LLC, Beverly Hills, California
  - Translational Clinical Research LLC, Aventura, Florida
  - Northwell Health, Great Neck, New York
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
- France (4):
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Claude Huriez, Lille
  - Hopital Europeen Marseille, Marseille
  - Hopital Pitie-Salpetriere, Paris
  - Centre Hospitalier Universitaire de Strasbourg - Nouvel hopital civil, Strasbourg
- Charite Universitätsmedizin Berlin, Berlin, Germany
- Poland (4):
  - Clinical Research Center Spzoo Medic-R Spolka Komandytowa, Poznan
  - Tomasz Blicharski Lubelskie Centrum Diagnostyczne, Świdnik
  - Medycyna Kliniczna Marzena Waszczak - Jeka, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 centers in the United States, France, and Poland from 10 April 2018 to 12 October 2021.
Pre-assignment Details: A total of 33 participants were randomized to AMG 592 or placebo in a 5:2 ratio (Cohorts 1, 2, and 3) or in a 1:3 ratio (Cohorts 4 and 5). Of those 33 participants, 2 were re-enrolled and re-randomized to subsequent cohorts upon completion. The total number of informed consent forms signed that led to randomization was 35.
Groups:
- Placebo: Matching placebo was administered by subcutaneous (SC) injection using dosing schedule A or B (A was less frequent than schedule B) for a total of 12 weeks.
  Two participants who completed Cohort 3 matching placebo dosing were subsequently re-enrolled in the study. One of the participants was randomized to matching placebo in Cohort 5. Participants re-enrolled to new cohorts were counted as different participants, as pre-specified.
- AMG 592 Cohort 1: A low dose of AMG 592 was administered by SC injection using dosing schedule A (less frequent than schedule B) for a total of 12 weeks.
- AMG 592 Cohort 2: A medium dose of AMG 592 was administered by SC injection using dosing schedule A (less frequent than schedule B) for a total of 12 weeks.
- AMG 592 Cohort 3: A medium dose of AMG 592 was administered by SC injection using dosing schedule B (more frequent than schedule A) for a total of 12 weeks.
- AMG 592 Cohort 4: A medium/high dose of AMG 592 was administered by SC injection using dosing schedule A (less frequent than schedule B) for a total of 12 weeks.
- AMG 592 Cohort 5: A high dose of AMG 592 was administered by SC injection using dosing schedule A (less frequent than schedule B) for a total of 12 weeks.
  Two participants who completed Cohort 3 matching placebo dosing were subsequently re-enrolled in the study. One of the participants was randomized to AMG 592 in Cohort 5. Participants re-enrolled to new cohorts were counted as different participants, as pre-specified.
Period: Overall Study
Arm/Group | Placebo | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5
Started | 10 | 5 | 5 | 7 | 4 | 4
Completed | 9 | 5 | 2 | 4 | 2 | 2
Not Completed | 1 | 0 | 3 | 3 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Decision by sponsor | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set: All participants who received at least 1 dose of investigational product. Participants re-enrolled to new cohorts were counted as different participants, as pre-specified.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5 | Total
Number analyzed (Participants) | 10 | 5 | 5 | 7 | 4 | 4 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (17.4) | 44.4 (13.4) | 44.4 (9.2) | 13.9 (63.0) | 16.6 (57.0) | 6.6 (60.0) | 14.4 (54.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 5 | 6 | 4 | 4 | 30
  Male | 2 | 2 | 0 | 1 | 0 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 5 | 5 | 7 | 4 | 4 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 0 | 0 | 3 | 3 | 2 | 12
  Black or African American and American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 4 | 5 | 5 | 4 | 1 | 2 | 21
  African and White | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Adverse Event (TEAE)
Description: A TEAE was defined as any adverse event (AE) starting on or after the first dose of investigational product through to the safety follow-up visit. Any clinically significant changes in physical examinations, vital signs, and clinical laboratory test results were recorded as AEs.
Time Frame: Day 1 up to end of study, maximum of 18 weeks (12-week double-blind treatment, 6-week safety follow-up)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5
Number analyzed (Participants) | 10 | 5 | 5 | 7 | 4 | 4
Participants | 7 | 5 | 5 | 7 | 3 | 4

2. Secondary Outcome: Maximum Observed Concentration (Cmax) for AMG 592
Time Frame: Day 1 (pre-dose) and 6 to 72 hours post-dose, and Days 8, 11, 15, 22, 29, 36, 43, 50, 57, 64, 71, 78, Day 85 (pre-dose) and 6 to 72 hours post-dose, and Days 92, 99, 113 and 127
Population: The Pharmacokinetic (PK) Parameter Analysis Set: All participants who have received AMG 592 and for whom at least one PK parameter could be adequately estimated. Only participants with PK data available for analysis are presented. Participants re-enrolled to new cohorts were counted as different participants, as pre-specified.
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5
Number analyzed (Participants) | 5 | 5 | 7 | 4 | 4
ng/mL
  First dose (Day 1) | 7.92 [5.52 to 13.8] | 13.0 [5.01 to 15.8] | 25.7 [9.74 to 43.7] | 30.7 [16.2 to 37.7] | 44.3 [29.6 to 67.9]
  Last dose (Day 85): number analyzed (Participants) | 5 | 2 | 2 | 2 | 2
  Last dose (Day 85) | 9.24 [7.05 to 13.7] | 18.9 [14.0 to 23.7] | 10.0 [8.77 to 11.3] | 56.5 [47.1 to 65.8] | 51.6 [25.7 to 77.5]

3. Secondary Outcome: Time of Cmax (Tmax) for AMG 592
Time Frame: as for outcome 2
Population: The PK Parameter Analysis Set: All participants who have received AMG 592 and for whom at least one PK parameter could be adequately estimated. Only participants with PK data available for analysis are presented. Participants re-enrolled to new cohorts were counted as different participants, as pre-specified.
Measure: Median (Full Range); unit: hours
Arm/Group | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5
Number analyzed (Participants) | 5 | 5 | 7 | 4 | 4
hours
  First dose (Day 1) | 24.0 [12.0 to 74.2] | 47.6 [20.3 to 48.0] | 24.1 [11.9 to 48.0] | 24.6 [24.0 to 27.1] | 17.8 [11.9 to 24.0]
  Last dose (Day 85): number analyzed (Participants) | 5 | 2 | 2 | 2 | 2
  Last dose (Day 85) | 25.2 [18.8 to 47.5] | 26.2 [23.4 to 28.9] | 18.0 [12.0 to 24.1] | 24.1 [23.5 to 24.7] | 16.7 [12.0 to 21.4]

4. Secondary Outcome: Area Under the Concentration-time Curve Over a Dosing Interval (AUCtau) for AMG 592
Time Frame: as for outcome 2
Population: as for outcome 3
Measure: Mean (Full Range); unit: hour*ng/mL
Arm/Group | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5
Number analyzed (Participants) | 5 | 4 | 4 | 2 | 3
hour*ng/mL
  First dose (Day 1) | 538 [261 to 986] | 915 [317 to 1360] | 1560 [971 to 2730] | 1960 [1960 to 1960] | 3770 [2020 to 5680]
  Last dose (Day 85): number analyzed (Participants) | 5 | 2 | 2 | 2 | 2
  Last dose (Day 85) | 773 [444 to 1160] | 1120 [779 to 1460] | 542 [347 to 736] | 3260 [2110 to 4420] | 3010 [1090 to 4930]

5. Secondary Outcome: Number of Participants With Anti-AMG 592 Binding Antibodies and Anti-Interleukin (IL-2) Binding Antibodies
Description: Number of participants who tested positive for developing anti-AMG 592 or anti-IL-2 binding antibodies at 1 or more post-baseline time points, with a negative or no result at baseline, are reported.
Time Frame: Day 1 up to end of study, maximum of 18 weeks (12-week double-blind treatment, 6-week safety follow-up)
Population: The Safety Analysis Set: All participants who received at least 1 dose of investigational product. Only participants who tested positive for anti-AMG 592 antibodies at anytime (pre- or post-dose) were analyzed for presence of anti-IL-2 neutralizing antibodies, as pre-specified. Participants re-enrolled to new cohorts were counted as different participants, as pre-specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5
Number analyzed (Participants) | 10 | 5 | 5 | 7 | 4 | 4
Participants
  Binding anti-AMG 592 antibody | 0 | 3 | 3 | 6 | 2 | 4
  Binding anti-IL-2 antibody: number analyzed (Participants) | 0 | 4 | 5 | 6 | 3 | 4
  Binding anti-IL-2 antibody |  | 1 | 2 | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Anti-AMG 592 Neutralizing Antibodies and Anti-IL-2 Neutralizing Antibodies
Description: Number of participants who tested positive for developing anti-AMG 592 or anti-IL-2 neutralizing antibodies at 1 or more post-baseline time points, with a negative or no result at baseline, are reported.
Time Frame: Day 1 up to end of study, maximum of 18 weeks (12-week double-blind treatment, 6-week safety follow-up)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5
Number analyzed (Participants) | 10 | 5 | 5 | 7 | 4 | 4
Participants
  Neutralizing anti-AMG 592 antibody | 0 | 0 | 2 | 1 | 0 | 2
  Neutralizing anti-IL-2 antibody: number analyzed (Participants) | 0 | 4 | 5 | 6 | 3 | 4
  Neutralizing anti-IL-2 antibody |  | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to end of study, maximum of 18 weeks (12-week double-blind treatment, 6-week safety follow-up)
Description: The Safety Analysis Set: All participants who received at least 1 dose of investigational product. Participants re-enrolled to new cohorts were counted as different participants, as pre-specified.
Arm/Group | Placebo | AMG 592 Cohort 1 | AMG 592 Cohort 2 | AMG 592 Cohort 3 | AMG 592 Cohort 4 | AMG 592 Cohort 5
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/5 | 0/5 | 0/7 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/5 | 1/5 | 0/7 | 0/4 | 1/4
Other Adverse Events (participants affected / at risk) | 7/10 | 5/5 | 5/5 | 7/7 | 3/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | AMG 592 Cohort 1 (N=5) | AMG 592 Cohort 2 (N=5) | AMG 592 Cohort 3 (N=7) | AMG 592 Cohort 4 (N=4) | AMG 592 Cohort 5 (N=4)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | AMG 592 Cohort 1 (N=5) | AMG 592 Cohort 2 (N=5) | AMG 592 Cohort 3 (N=7) | AMG 592 Cohort 4 (N=4) | AMG 592 Cohort 5 (N=4)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Corneal opacity (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Reflux gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Administration site joint erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Administration site joint pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Administration site pruritus (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Administration site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Administration site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Application site joint swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cyst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 3 | 3 | 5 | 2 | 2
Injection site induration (General disorders) | 0 | 0 | 1 | 1 | 2 | 2
Injection site inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site mass (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Injection site pruritus (General disorders) | 0 | 1 | 1 | 2 | 2 | 2
Injection site rash (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 2 | 3 | 2 | 2 | 3
Injection site swelling (General disorders) | 0 | 0 | 0 | 1 | 1 | 1
Injection site warmth (General disorders) | 0 | 1 | 0 | 1 | 1 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 2 | 0 | 0 | 0
Urethritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/22/NCT03451422/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT03451422/SAP_001.pdf